CLINICAL TRIAL: NCT01443208
Title: A Phase 1, Randomized, Subject- and Investigator-Blind, Placebo-Controlled, Parallel-Group, Single and Multiple-Dose Study of Desvenlafaxine in Korean Healthy Subjects
Brief Title: Pharmacokinetics and Safety of Desvenlafaxine in Korean Healthy Subjects Following Single and Multiple Oral Doses of Desvenlafaxine Succinate Sustained Release Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: B2061137
Record Dates: First submitted 2011-09-23; First posted 2011-09-29 (Estimated); Last update posted 2012-01-02 (Estimated); Status verified 2011-12

CONDITIONS: Major Depressive Disorder
Keywords: pharmacokinetics; safety; desvenlafaxine; Korean healthy subjects
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 50 mg (Experimental)
  Interventions: Drug: desvenlafaxine
- 100 mg (Experimental)
  Interventions: Drug: desvenlafaxine
- 200 mg (Experimental)
  Interventions: Drug: desvenlafaxine

INTERVENTIONS:
Drug: desvenlafaxine — one 50 mg desvenlafaxine succinate sustained-release tablet or matching placebo, single dose and once daily dose for 5 days
  Arms: 50 mg
Drug: desvenlafaxine — one 100 mg desvenlafaxine succinate sustained-release tablet or matching placebo, single dose and once daily dose for 5 days
  Arms: 100 mg
Drug: desvenlafaxine — two 100 mg desvenlafaxine succinate sustained-release tablets or matching placebo, single dose and once daily dose for 5 days
  Arms: 200 mg

SUMMARY:
To evaluate the pharmacokinetics and safety of single dose and multiple doses of desvenlafaxine in Korean healthy subjects and compare to westerners.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects
* Between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs)

Exclusion Criteria:

* Elevated risk of suicide, in the opinion of the investigator or expert consultant
* Pregnant or nursing females
* Females of childbearing potential who are unwilling or unable to use an acceptable method of contraception

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
For single dose: maximum concentration (Cmax) | day 1
For single dose: time to first occurence of Cmax (Tmax) | day 1
For single dose: area under curve (0-time for last quantifiable concentration) (AUClast) | day 1
For multiple dose: maximum concentration (Cmax) | day 8
For multiple dose: time to first occurence of Cmax (Tmax) | day 8
For multiple dose: trough concentration (Ctrough) | day 8
For multiple dose: area under curve (0-24hours) (AUC0-24) | day 8

SECONDARY OUTCOMES:
For single dose if data permit: terminal elimination half life (t1/2) | day 1
For single dose if data permit: area under curve (0-infinity) (AUCinf) | day 1
For single dose if data permit: oral clearance (CL/F) | day 1
For single dose if data permit: apparent volume of distribution (Vz/F) | day 1
For multiple dose if data permit: accumulation factor (Rac) | day 8
For multiple dose if data permit: terminal elimination half life (t1/2) | day 8
For multiple dose if data permit: oral clearance (CL/F) | day 8
For multiple dose if data permit: apparent volume of distribution (Vz/F) | day 8

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Seoul, South Korea

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2061137&StudyName=Pharmacokinetics%20and%20Safety%20of%20Desvenlafaxine%20in%20Korean%20Healthy%20Subjects%20Following%20Single%20and%20Multiple%20Oral%20Doses%20of%20Desvenlafaxine%20Succinat